CLINICAL TRIAL: NCT04531241
Title: Clinical Evaluation of Senofilcon A Contact Lenses Using a Novel Manufacturing Technology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johnson & Johnson Vision Care, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR-6417
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Results first posted 2021-12-14 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-11

CONDITIONS: Visual Acuity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Test/Control (Experimental): Eligible subjects that are habitual wearers of daily disposable contact lenses in both eyes will be randomly assigned to sequence, Test/Control.
  Interventions: Device: ACUVUE® OASYS 1-DAY
- Control/Test (Experimental): Eligible subjects that are habitual wearers of daily disposable contact lenses in both eyes will be randomly assigned to sequence, Control/Test.
  Interventions: Device: ACUVUE® OASYS 1-DAY

INTERVENTIONS:
Device: ACUVUE® OASYS 1-DAY — senofilcon A contact lenses made with a novel manufacturing technology
  Other Names: TEST
Device: ACUVUE® OASYS 1-DAY — senofilcon A contact lenses made with the current manufacturing technology
  Other Names: CONTROL

SUMMARY:
This study is a multi-site, randomized, double-masked, 2×2 crossover design, 1-week dispensing study. Subjects will wear bilaterally both Test and Control lenses in a random order for 1-week each as a daily disposable modality with a wash-out period of 1 week between the wearing periods.

ELIGIBILITY:
Inclusion Criteria:

1. The subject must read, understand, and sign the STATEMENT OF INFORMED CONSENT and receive a fully executed copy of the form.
2. Appear able and willing to adhere to the instructions set forth in this clinical protocol.
3. Must be at least 18 and not more than 70 years of age (including 70) at the time of screening.
4. The subject must be a habitual and adapted wearer of daily disposable contact lenses in both eyes (at least 1 month of daily wear).
5. The subject must have normal eyes (i.e., no ocular medications or infections of any type).
6. The subject's required spherical contact lens prescription must be in the range of -0.50 to -3.25 and -3.75 to -6.00 D in each eye.
7. The subject's refractive cylinder must be ≤0.75D in each eye, if present
8. The subject must have best corrected visual acuity of 20/25 or better in each eye.

Exclusion Criteria:

1. Currently pregnant or lactating (subjects who become pregnant during the study will be discontinued).
2. Any systemic disease, autoimmune disease, or use of medication that may interfere with contact lens wear. (at the discretion of the investigator)
3. Any previous, or planned, ocular or interocular surgery (e.g., radial keratotomy, PRK, LASIK, etc.).
4. Any ocular infection.
5. Any corneal distortion resulting from previous hard or rigid gas permeable contact lens wear.
6. Monovision or multi-focal contact lens correction.
7. Participation in any contact lens or lens care product clinical trial within 7 days prior to study enrollment.
8. History of binocular vision abnormality or strabismus.
9. Any infectious disease (e.g., hepatitis, tuberculosis) or a contagious immunosuppressive disease (e.g., HIV, by self-report).
10. Suspicion of or recent history of alcohol or substance abuse.
11. History of serious mental illness.
12. History of seizures.
13. Employee or immediate family member of an employee of clinical site (e.g., Investigator, Coordinator, Technician)
14. Any ocular allergies, infections or other ocular abnormalities that are known to interfere with contact lens wear and/or participation in the study. This may include, but not be limited to entropion, ectropion, extrusions, chalazia, recurrent styes, glaucoma, history of recurrent corneal erosions, aphakia, or corneal distortion
15. Any Grade 3 or greater slit lamp findings (e.g., edema, corneal neovascularization, corneal staining, tarsal abnormalities, conjunctival injection) on the Food and Drug Administration (FDA) classification scale.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2020-09-25 (Actual); Study Completion 2020-09-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Vision Care, Inc. Clinical Trial, Study Director — Johnson & Johnson Vision Care, Inc.
Locations (7):
- United States (7):
  - Vue Optical Boutique, Jacksonville, Florida
  - Maitland Vision Center, Maitland, Florida
  - Tallahassee Eye Center, Tallahassee, Florida
  - VisionPoint Eye Center, Bloomington, Illinois
  - ProCare Vision Centers, Granville, Ohio
  - EyeCare Professionals of Powell, Powell, Ohio
  - Frazier Vision, Inc., Tyler, Texas

IPD SHARING:
Plan to Share IPD: Yes
Johnson & Johnson Medical Device Companies have an agreement with the Yale Open Data Access (YODA) to serve as the independent review panel for evaluation of requests for clinical study reports and participant level data from investigators and physicians for scientific research that will advance medical knowledge and public health. Requests for access to the study data can be submitted through the YODA Project site at http://yoda.yale.edu
URL: http://yoda.yale.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 136 subjects were enrolled in this study. Of those enrolled, 135 were dispensed at least one study lens while, 1 subject failed to meet all eligibility criteria. Of those subjects dispensed a study lens, 127 completed the study while, 8 subjects were discontinued from the study.
Groups:
- Senofilcon A (Test)/ Senofilcon A (Control): subjects that wore the senofilcon A (Test) lens in period 1 and the senofilcon A (Control) in period 2.
- Senofilcon A (Control)/ Senofilcon A (Test): subjects that wore the senofilcon A (Control) lens in period 1 and the senofilcon A (Test) in period 2.
Period: Period 1
Arm/Group | Senofilcon A (Test)/ Senofilcon A (Control) | Senofilcon A (Control)/ Senofilcon A (Test)
Started | 68 | 67
Completed | 64 | 65
Not Completed | 4 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Dispesed incorrect lens power | 1 | 0
Not completed — Protocol Violation | 1 | 0
Not completed — No longer eligible | 0 | 1
Not completed — Lens Discomfort | 0 | 1
Period: Period 2
Arm/Group | Senofilcon A (Test)/ Senofilcon A (Control) | Senofilcon A (Control)/ Senofilcon A (Test)
Started | 64 | 65
Completed | 63 | 64
Not Completed | 1 | 1
Not completed — Covid-19 Related | 1 | 1

BASELINE CHARACTERISTICS:
Population: All subjects dispensed a study lens.
Groups:
- Dispensed Subjects: All subjects dispensed a study lens.
Arm/Group | Dispensed Subjects
Number analyzed (Participants) | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (7.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94
  Male | 41
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 5
  Black or African American | 2
  White | 128
Region of Enrollment [Number; unit: participants]
  United States | 135

OUTCOME MEASURES:

1. Primary Outcome: Overall CLUE Comfort
Description: Overall comfort was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 1-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: unit on a scale
Groups:
- Senofilcon A (Test): Subjects that wore the Test lens in either the first or second period of the study.
- Senofilcon A (Control): Subjects that wore the Control lens in either the first or second period of the study.
Arm/Group | Senofilcon A (Test) | Senofilcon A (Control)
Number analyzed (Participants) | 108 | 108
unit on a scale | 60.9 (22.67) | 65.1 (21.47)
Statistical Analysis 1: Comparison: Senofilcon A (Test) vs Senofilcon A (Control); Test type: Non-Inferiority — It was calculated that 120 participants randomized in a 1:1 fashion between the two sequences would have at least 80% power to detect a 5 points difference in mean overall comfort and vision at the 1-week follow-up. Sample size was determined using Stroup's Method (alpha=0.05). A non-inferiority margin of -5 points was used; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-Square Mean Difference = -2.9, 95% CI 2-sided [-6.8 to 1.1], Standard Error of Mean 2.01 — Mean difference was calculated as Test - Control

2. Secondary Outcome: Visual Performance
Description: Visual performance was calculated as monocular contact lens-corrected distance visual acuity using a logMAR visual acuity scale. This was evaluated under both high luminance/low contrast conditions and low luminance/high contrast conditions at 4 meters from Early Treatment Diabetic Retinopathy Study (ETDRS) charts. The room illuminance was required to be between 7.3 and 7.9 EV (394-597 lux). For high illumination, the room was required to be >400 lux with low contrast charts. For low illumination, the room was required to be <2.5 lux. Letter-by-letter results calculated the visual performance score for each chart read. logMAR scores closer to zero, or below zero, indicate a better visual acuity. A logMAR visual performance score of 0.0 is equivalent to Snellen visual acuity of 20/20.
Time Frame: 1-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | Senofilcon A (Test) | Senofilcon A (Control)
Number analyzed (Participants) | 108 | 108
logMAR
  Under Low Luminance High Contrast Condition | 0.02 (0.092) | 0.03 (0.094)
  Under High Luminance Low Contrast Condition | 0.02 (0.101) | 0.03 (0.093)
Statistical Analysis 1: Comparison: Senofilcon A (Test) vs Senofilcon A (Control); Low Luminance High Contrast; Test type: Non-Inferiority — It was calculated that 120 participants randomized in a 1:1 fashion between the two sequences would have a 0.05 logMAR unit difference in logMAR visual acuity at LLHC and HLLC lighting conditions at the 1-week follow-up. Sample size was determined using Stroup's Method (alpha=0.05). A non-inferiority margin of 0.05 logMAR units was used; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-Square Mean Difference = -0.010, 95% CI 2-sided [-0.0199 to 0.0], Standard Error of Mean 0.0050 — Mean difference was calculated as Test - Control
Statistical Analysis 2: Comparison: Senofilcon A (Test) vs Senofilcon A (Control); High Luminance Low Contrast; Test type: Non-Inferiority — [test comment as in outcome 2, analysis 1]; Mixed Model Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-Square Mean Difference = -0.004, 95% CI 2-sided [-0.0173 to 0.0087], Standard Error of Mean 0.0066 — Mean difference was calculated as Test - Control

3. Secondary Outcome: Average Daily Wear Time (in Hours)
Description: Average daily wear time was calculated as the number of hours between subjects reported time of insertion and time of removal of the study lenses, on an average day, at 1-Week Follow up evaluation.
Time Frame: 1-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Senofilcon A (Test) | Senofilcon A (Control)
Number analyzed (Participants) | 108 | 108
hours | 14.3 (1.93) | 14.4 (1.90)
Statistical Analysis 1: Comparison: Senofilcon A (Test) vs Senofilcon A (Control); Test type: Non-Inferiority — It was calculated that 120 participants randomized in a 1:1 fashion between the two sequences would have a 1 hour difference in average daily wear time at the 1-week follow-up. Sample size was determined using Stroup's Method (alpha=0.05). A non-inferiority margin of 1 hour was used; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-Square Mean Difference = -0.052, 95% CI 2-sided [-0.1968 to 0.0933], Standard Error of Mean 0.0731 — Mean difference was calculated as Test - Control

4. Primary Outcome: Overall CLUE Vision
Description: Overall vision was assessed using the Contact Lens User Experience™ (CLUE) questionnaire. CLUE is a validated patient-reported outcomes (PRO) questionnaire to assess patient experience attributes of soft contact lenses (comfort, vision, handling, and packaging) in a contact-lens wearing population in the US, ages 18-65. Derived CLUE scores using Item Response Theory (IRT) follow a normal distribution with a population average score of 60 (SD 20), where higher scores indicate a more favorable/positive response with a range of 0-120.
Time Frame: 1-Week Follow-up
Population: Subjects that completed all study visits without a major protocol deviation.
Measure: Mean (Standard Deviation); unit: unit on a scale
Arm/Group | Senofilcon A (Test) | Senofilcon A (Control)
Number analyzed (Participants) | 108 | 108
unit on a scale | 65.5 (19.31) | 67.8 (17.79)
Statistical Analysis 1: Comparison: Senofilcon A (Test) vs Senofilcon A (Control); Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Mixed Models Analysis; Linear mixed model using the Kenward and Roger method for the denominator degrees of freedom; Least-Square Mean Difference = -2.6, 95% CI 2-sided [-5.5 to 0.3], Standard Error of Mean 1.47 — Mean difference was calculated as Test - Control

ADVERSE EVENTS:
Time Frame: Throughout the duration of the study; approximately 1 month per subject.
Arm/Group | Senofilcon A (Test) | Senofilcon A (Control)
All-Cause Mortality (participants affected / at risk) | 0/135 | 0/135
Serious Adverse Events (participants affected / at risk) | 0/135 | 0/135
Other Adverse Events (participants affected / at risk) | 0/135 | 0/135

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-10): https://cdn.clinicaltrials.gov/large-docs/41/NCT04531241/Prot_SAP_000.pdf